CLINICAL TRIAL: NCT00196872
Title: A Phase III Trial to Compare ETC vs, EC-TX and Ibandronate vs. Observation in Patients With Node-positive Primary Breast Cancer (GAIN)
Brief Title: A Study to Compare ETC vs. EC-TX and Ibandronate vs. Observation in Patients With Node-positive Primary Breast Cancer (GAIN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GBG 33; GAIN
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: dose dense sequence; dose dense combination; node positive disease
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Paclitaxel; Capecitabine

ARMS (4):
- ETC-with Ibandronat (Experimental): ETC follwoed by Ibandronat
  Interventions: Drug: Epirubicine; Drug: Cyclophosphamide; Drug: Taxol; Drug: Ibandronat
- ETC without Ibandronat (Experimental): ETC not followed by Ibandronat
  Interventions: Drug: Epirubicine; Drug: Cyclophosphamide; Drug: Taxol
- EC-TX with Ibandronat (Experimental): EC-TX followed by Ibandronat
  Interventions: Drug: Epirubicine; Drug: Cyclophosphamide; Drug: Taxol; Drug: Xeloda; Drug: Ibandronat
- EC-TX without Ibandronat (Experimental): EC-TX not followed by Ibandronat
  Interventions: Drug: Epirubicine; Drug: Cyclophosphamide; Drug: Taxol; Drug: Xeloda

INTERVENTIONS:
Drug: Epirubicine — Epirbubicne is given
Drug: Cyclophosphamide — Cyclophosphamide is given
Drug: Taxol — Taxol is given
Drug: Xeloda — Xeloda is given
  Arms: EC-TX with Ibandronat; EC-TX without Ibandronat
Drug: Ibandronat — Ibandronat is given
  Arms: EC-TX with Ibandronat; ETC-with Ibandronat

SUMMARY:
In the recent AGO-study, a dose-dense and dose-intensified sequence of Epirubicin - Paclitaxel - Cyclophosphamide has shown superior efficacy compared to a conventionally dosed sequence of Epirubicin / Cyclophosphamid and Paclitaxel and was therefore chosen as standard treatment in this study.

The experimental arm of EC-TX combines several strategies: the combination of EC will be administered every 2 weeks as a dose-dense regimen, the combination of TX can also be considered as dose-dense due to the weekly application of paclitaxel. Furthermore there is clinical evidence, that a combination of capecitabine and Paclitaxel provide synergistic effects with improved tumour response. A randomized phase III study could demonstrate a survival benefit of a combination of capecitabine with Docetaxel in patients with metastatic breast cancer. This synergistic effect is probably based on the preclinical observed taxane-mediated up-regulation of thymidine phosphorylase in the tumour cell, which give drive to an increased transformation of capecitabine to its active form 5-Fluorouracil. Apart from this synergy, the EC-TX regimen includes now 4 highly active compounds for the treatment of breast cancer. The total doses of Epirubicin and Paclitaxel are identical in both arms. The dosage of Cyclophosphamide is lower in the experimental arm, which is preferred due to the induction of leukaemia at higher doses of Cyclophosphamide. The duration of both arms with 18 and 20 weeks is nearly similar.

The 2 by 2 factorial design of the trial provides the additional possibility to explore the efficacy of a bisphosphonate as another strategy to further improve the prognosis of node positive breast cancer.

DETAILED DESCRIPTION:
Currently several strategies are under investigation to further improve adjuvant treatment of early node-positive breast cancer. These are combination treatment of drugs with synergistic mode of action, dose-dense application of cytotoxic drugs, dose-intensification and the use of new, non-cytotoxic approaches.

In the recent AGO-study, a dose-dense and dose-intensified sequence of Epirubicin - Paclitaxel - Cyclophosphamide has shown superior efficacy compared to a conventionally dosed sequence of Epirubicin / Cyclophosphamid and Paclitaxel and was therefore chosen as standard treatment in this study.

The experimental arm of EC-TX combines several of the above mentioned strategies: the combination of EC will be administered every 2 weeks as a dose-dense regimen, the combination of TX can also be considered as dose-dense due to the weekly application of paclitaxel. Furthermore there is clinical evidence, that a combination of capecitabine and Paclitaxel provide synergistic effects with improved tumour response. A randomized phase III study could demonstrate a survival benefit of a combination of capecitabine with Docetaxel in patients with metastatic breast cancer. This synergistic effect is probably based on the preclinical observed taxane-mediated up-regulation of thymidine phosphorylase in the tumour cell, which give drive to an increased transformation of capecitabine to its active form 5-Fluorouracil. Apart from this synergy, the EC-TX regimen includes now 4 highly active compounds for the treatment of breast cancer. The total doses of Epirubicin and Paclitaxel are identical in both arms. The dosage of Cyclophosphamide is lower in the experimental arm, which is preferred due to the induction of leukaemia at higher doses of Cyclophosphamide. The duration of both arms with 18 and 20 weeks is nearly similar.

The 2 by 2 factorial design of the trial provides the additional possibility to explore the efficacy of a bisphosphonate as another strategy to further improve the prognosis of node positive breast cancer. As the mechanism of action of cytotoxic drugs and bisphosphonates appear to be independent the factorial design is an adequate statistical model for this trial. Up to now only limited information is available on the potential role of bisphosphonates in this setting and they have all been generated by using the 1st generation bisphosphonate Clodronate. 3rd generation bisphosphonates like ibandronate are much more active, less toxic and their application is more convenient (which is of high importance regarding the long duration of treatment).

Primary aims of this trial are to improve disease-free survival by using the EC-TX regimen and by using ibandronate as adjuvant treatment for 2 years.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements, Histologically confirmed unilateral or bilateral primary carcinoma of the breast Age at diagnosis at least 18 years and biologically younger than 65 years Adequate surgical treatment with histological complete resection (R0) of the tumor and at least 10 axillary nodes At least one histological involved axillary or internal mammarian lymph node No evidence for distant metastasis after complete diagnostic work up Primary wound healing from breast surgery without signs of infection Performance Status ECOG < 2 Estimated life expectancy of at least 10 years irrespective of the diagnosis of breast cancer The patient must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating center which could be the Principal or an Co- investigator's site

Exclusion Criteria:

Known hypersensitivity reaction to the compounds or incorporated substances or known dihydropyrimidine dehydrogenase (DHP) deficiency.

Inadequate organ function including: ANC < 1.5 G/l, Platelets < 100 G/l , Transaminases, Creatinine or Bilirubin > 1.25 times above upper normal limits (UNL), AP > 3 times above UNL, Creatinine Clearance < 30ml/min (if Creatinine is above UNL, according to Cockroft-Gault), severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study Insufficient and uncompensated cardiac function with LVEF below the normal range of the institution, history of severe heart disease, myocardial infarction within the last 6 months, cardiac arrhythmias LOWN II Evidence for infection including wound infections, HIV, Hepatitis Secondary malignancy, except curatively treated basalioma of the skin and carcinoma in situ of the cervix Time since axillary dissection > 3 months (optimal < 1 month) Non-operable breast cancer Previous and already (neoadjuvant or adjuvant) treated invasive breast carcinoma Previous or concurrent anti-tumor treatment for any reason Simultaneous therapy with Sorivudine or Brivudine as virostatics, immunosuppressive treatment or concurrent treatment with aminoglycosides Pregnancy or lactation period. Adequate non hormonal contraception is a prerequisite in premenopausal patients Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.

Male patients

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2004-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
A: To compare the disease-free survival after adjuvant chemotherapy with "ETC" (Arm A1) or "EC-TX" (Arm A2) in patients with primary node-positive breast cancer. | US-law not applicable
B: To compare the disease-free survival with (Arm B1) or without ibandronate (Arm B2) treatment for 2 years in patients with primary node-positive breast cancer | US-law not applicable

SECONDARY OUTCOMES:
To compare overall survival between arms A1 vs. A2 and B1 vs. B2 | US-law not applicable
To evaluate the compliance in arms A1 vs. A2 and in B1 | US-law not applicable
To compare the safety between arms A1 vs. A2 and B1 vs. B2 | US-law not applicable
To assess the rate of responders to erythropoesis stimulating factors in arm A1 and A2 | US-law not applicable
To compare the incidence of secondary primaries between arms A1 vs. A2 | US-law not applicable
To compare the event-free survival in subgroups of hormone sensitive and insensitive disease and in groups with 1-3, 4-9 or 10+ involved nodes between arms A1 vs. A2 and B1 vs. B2 | US-law not applicable
Tertiary objectives: | US-law not applicable
To determine prognostic factors like TS or TP and others on tumor tissue collected from primary surgery and to correlate them with study treatment effect | US-law not applicable

CONTACTS AND LOCATIONS:
Overall Officials: Volker Möbus, Prof. Dr., Principal Investigator — Städtische Kliniken Frankfurt a.M.-Höchst, Gotenstr. 6-8, 65929 Frankfurt, Germany
Locations (1):
- Städtische Kliniken Frankfurt a.M.-Höchst, Frankfurt, Hessia, Germany

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Sturken C, Mobus V, Milde-Langosch K, Schmatloch S, Fasching PA, Ruschoff J, Stickeler E, Henke RP, Denkert C, Hanker L, Schem C, Vladimirova V, Karn T, Nekljudova V, Kohne CH, Marme F, Schumacher U, Loibl S, Muller V. TGFB-induced factor homeobox 1 (TGIF) expression in breast cancer. BMC Cancer. 2021 Aug 14;21(1):920. doi: 10.1186/s12885-021-08656-0. PMID 34391399
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Noske A, Mobus V, Weber K, Schmatloch S, Weichert W, Kohne CH, Solbach C, Ingold Heppner B, Steiger K, Muller V, Fasching P, Karn T, van Mackelenbergh M, Marme F, Schmitt WD, Schem C, Stickeler E, Loibl S, Denkert C. Relevance of tumour-infiltrating lymphocytes, PD-1 and PD-L1 in patients with high-risk, nodal-metastasised breast cancer of the German Adjuvant Intergroup Node-positive study. Eur J Cancer. 2019 Jun;114:76-88. doi: 10.1016/j.ejca.2019.04.010. Epub 2019 May 7. PMID 31075727
- See also: Related Info — http://www.germanbreastgroup.de